CLINICAL TRIAL: NCT04874831
Title: A Phase II, Open Label, Multicenter Study to Investigate the Efficacy and Safety of Domatinostat in Combination With Avelumab in Patients With Treatment-naïve Metastatic Merkel Cell Carcinoma - the MERKLIN 1 Study
Brief Title: Domatinostat in Combination With Avelumab in Patients With Treatment-naïve Metastatic Merkel Cell Carcinoma (MERKLIN 1)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Refocusing of sponsor's clinical development program. No safety concern or change of the risk-benefit assessment of the investigational medicinal product has led to this decision.
Sponsor: 4SC AG (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-202-4-2019; 2019-003575-19 (EudraCT Number)
Record Dates: First submitted 2021-04-15; First posted 2021-05-06 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — domatinostat; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- domatinostat and avelumab (Experimental): Single arm study of Domatinostat tablets in combination with avelumab infusion
  Interventions: Drug: domatinostat in combination with avelumab

INTERVENTIONS:
Drug: domatinostat in combination with avelumab — domatinostat tablets and avelumab infusion

SUMMARY:
This phase II trial studies how well domatinostat (4SC-202) works in combination with avelumab in adult patients with treatment-naïve metastatic Merkel Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age 18 years at signature of Informed Consent Form (ICF).
3. Histologically proven MCC.

   * Confirmation of the diagnosis by immune-histochemistry as per standard at the institution, including (but not limited to) CK20 and TTF-1.
   * Patients must have metastatic or distally recurrent disease; Ml status must be confirmed at entry.
   * Patients must not have received any prior systemic treatment for metastatic MCC. Prior treatment in the adjuvant setting (no clinically detectable disease; no metastatic disease) will be allowed, if the end of the treatment occurred at least 6 months prior to study entry, i.e. signing ICF.
4. Fresh biopsy or archival tumor tissue (not older than 3 months) from an unirradiated lesion.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at study entry.
6. Estimated life expectancy of more than 12 weeks.
7. Disease must be measurable with at least one unidimensional measurable lesion by RECIST vl.l (including skin lesions).
8. Adequate hematological and organ function defined by the following parameters:

   Adequate hematological function defined by
   * White blood cell count (WBC) > 3000/pl
   * Absolute Neutrophil Count (ANC) > 1500/pl
   * Lymphocyte count > 500/pl
   * Hemoglobin (Hb) > 9 g/dl (or > 5.6 mmol/L), may have been transfused
   * Platelet count > 100.000/pl

   Adequate hepatic function defined by
   * Serum total bilirubin < 1.5 x ULN
   * ALT and/or AST < 1.5 x ULN

   Adequate renal function defined by

   • eGFR > 60 ml/ min (as per Cockcroft-Gault formula)
9. Highly effective contraception for both male and female subjects if the risk of conception exists. Female patients of childbearing potential must have a negative urine or serum pregnancy test before receiving the first dose of study medication and must comply with contraception methods as requested by the study protocol.

Exclusion Criteria:

1. Participation in another interventional clinical study within the past 30 days (participation in observational studies is permitted)
2. Concurrent treatment with a non-permitted drug.
3. Prior therapy with any histone deacetylase (HDAC) inhibitor or antibody/drug targeting T cell coregulatory proteins (immune checkpoints) such as anti-programmed death 1 (PD-1), antiprogrammed death-ligand 1 (PD-L1) or anti-cytotoxic T-lymphocyte antigen-4 (CTLA-4) antibody.
4. Concurrent anti-cancer treatment (for example, cytoreductive therapy, radiotherapy, immune therapy, or cytokine therapy except for erythropoietin). Radiotherapy administered to superficial lesions is not allowed if such lesions are considered target lesions in the efficacy evaluation or may influence the efficacy evaluation of the study treatment.
5. Major surgery for any reason, except diagnostic biopsy, within 4 weeks and/or if the subject has not fully recovered from surgery.
6. Concurrent systemic therapy with steroids or other immunosuppressive agents (e.g. methotrexate, azathioprine, interferons, mycophenolate, anti-TNF agents and other), or the use of any investigational drug within 28 days before the start of study treatment. Short-term administration of systemic steroids e.g. for allergic reactions or the management of immune-related adverse events [irAE] while on study is allowed. Also, patients requiring hormone replacement with corticosteroids for adrenal insufficiency are eligible if the steroids are administered only for purpose of hormonal replacement and at doses < 10 mg or equivalent prednisone per day.
7. Conditions requiring systemic anti-arrhythmic therapy known to prolong QT/QTc interval, patients with QTcF interval >480 msec on at least 2 separate and consecutive ECGs at screening or a medical history of long-QT-Syndrome.
8. Patients with active central nervous system (CNS) metastases are excluded and a brain CT/MRI will be required during screening if not performed within 6 weeks prior to the planned start of the study treatment. Subjects with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy.
9. History of or concurrent malignancies, except the malignancy is clinically insignificant, no systemic treatment is or has been required for the last 6 months, and the patient is clinically stable
10. Prior organ transplantation (including allogeneic stem-cell transplantation).
11. Any active gastrointestinal disorder that could interfere with the absorption of domatinostat characterized by malabsorption or inability to swallow tablets as per judgment of the Investigator.
12. Positive testing for HIV or known AIDS or HBV or HCV infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening is positive).
13. Active or history of any autoimmune disease (except for patients with vitiligo) or immune-diseases that required treatment with systemic immune modulating drugs.
14. History or current evidence of clinically relevant allergies or hypersensitivity, which includes known or suspected intolerabilities attributed to domatinostat or avelumab or to constituents of the domatinostat tablets or avelumab infusion and known severe hypersensitivity reactions (Grade 3) to monoclonal antibodies.
15. Persisting toxicity related to prior therapy Grade > 1 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0; however, sensory neuropathy Grade < 2 will be acceptable.
16. Pregnancy or lactation period.
17. Known or suspected alcohol or drug abuse.
18. Clinically significant (i.e. active) cardiovascular and/or thromboembolic diseases:

    * Cerebral vascular accident or stroke < 6 months prior to enrollment.
    * Uncontrolled hypertension
    * Congestive heart failure (New York Heart Association (NYHA) ClassIII or IV)
    * Serious cardiac arrhythmia requiring medication (patients with status post pacemaker and/or defibrillator implantation can be included)
    * Symptomatic ischemic or severe valvular heart disease
    * Unstable angina pectoris or a myocardial infarction within 6 months prior to screening, i.e. signing ICF
19. All other significant diseases (for example, inflammatory bowel disease), which, in the opinion of the Investigator, might impair the patient s tolerance to the study treatment.
20. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
21. Legal incapacity or limited legal capacity.
22. Administration of a live vaccine within 28 days prior to study drug administration. Live vaccines are also prohibited during study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response (OR) | up to 1 year
  Confirmed Objective Response (OR) according to RECIST vl.l, determined by independent review. Both Complete Response and Partial Response must be confirmed by a second tumor assessment preferably at the regularly scheduled 6-weeks assessment interval, but no sooner than 4 weeks after the initial diagnosis of CR or PR.

SECONDARY OUTCOMES:
Duration of Response (DOR) | up to 1 year
  Duration of Response (DOR) according to RECIST vl.l as determined by independent review.
Durable Response (DR) | up to 1 year
  Durable Response (DR) according to RECIST vl.l, defined as objective response (CR or PR) determined by independent review with duration of at least 6 months.
Overall Survival (OS) | approx 3.5 years
  Overall Survival (OS) time, defined as the time from the first administration of study treatment until death due to any cause determined by the Investigator.
Progression Free Survival (PFS) | approx. 3 years
  Progression Free Survival (PFS) according to RECIST vl.l, defined as the time from first dosing (Day 1) to the date of PD or death from any cause (whichever comes first) as determined by independent review.
Disease Control (DC) | up to 1 year
  Disease Control (DC) according to RECIST vl.l, defined as the proportion of patients with either an objective response (CR, PR) or stable disease (SD), as determined by independent review.
RECIST vl.l response | up to 1 year
  RECIST vl.l responses at 6 and 12 months after start of study treatment as determined by independent review.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | approx. 3 years
  number, frequency, duration and severity of AEs
Correlation of biomarker expression to efficacy | up to 1 year
  Correlation of ORR, DOR, DR, DC and PFS to biomarker expression determined by immunohistochemistry.
Anti-drug-antibodies (ADAs) | up to 1 year
  Anti-drug-antibodies (ADAs) treatments.
Health related Quality of Life determined by the questionnaire FACT-M | up to 1 year
  The impact of treatment on the patient's QoLwill be assessed with the questionnaire "Functional Assessment of Cancer Therapy - Melanoma (FACT-M)" where QoL is assessed on a scale 0-240 (higher score means better status of health)
Plasma concentration of domatinostat and avelumab | up to 1 year
  Single trough values of domatinostat and avelumab at pre-defined time points
Health related Quality of Life determined by the questionnaire EQ-5D-5L | up to 1 year
  The impact of treatment on the patient's QoLwill be assessed with the questionnaire "EQ-5D-5L" which is a multi attribute utility instrument for measuring health-related QoL as EQ5D index with a score 0-1 (higher score means better status of health)

IPD SHARING:
Plan to Share IPD: No